CLINICAL TRIAL: NCT06531369
Title: Application of Flumazenil to Antagonize Remimazolam and Evaluation of Remimazolam Plasma Concentration in Kidney Transplant Patients: A Randomized Controlled Trial
Brief Title: Flumazenil Antagonism of Remimazolam in Kidney Transplant Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Wu, Chief Physician, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YXLL-KY-2024(059)
Record Dates: First submitted 2024-06-22; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Flumazenil to Antagonize Remimazolam; Remimazolam; Renal Transplantation
Keywords: Flumazenil; Remimazolam; renal transplantation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Flumazenil group 1（F1 group）"+"Flumazenil group 2（F2 group）" (Active Comparator): "Flumazenil group 1（F1）":Immediately after surgery, 0.5 mg flumazenil was administered, followed by an equal volume of saline (equal to the volume of 0.3 mg flumazenil) 25 minutes later.
  "Flumazenil group 2（F2）":Immediately after surgery, 0.5 mg flumazenil was administered, followed by 0.3 mg flumazenil 25 minutes later.
  Interventions: Drug: Flumazenil Injection（F1 group）; Drug: Flumazenil Injection（F2 group）
- Control Group (C group) (Placebo Comparator): Immediately after surgery, an equal volume of saline (equal to the volume of 0.5 mg flumazenil) was administered, followed by an equal volume of saline (equal to the volume of 0.3 mg flumazenil) 25 minutes later.
  Interventions: Drug: Saline（C group）

INTERVENTIONS:
Drug: Flumazenil Injection（F1 group） — Flumazenil Injection（F1 group）: Immediately after surgery, 0.5 mg flumazenil was administered, followed by an equal volume of saline (equal to the volume of 0.3 mg flumazenil) 25 minutes later.
  Other Names: Flumazenil at Different Dosages
  Arms: "Flumazenil group 1（F1 group）"+"Flumazenil group 2（F2 group）"
Drug: Flumazenil Injection（F2 group） — Flumazenil Injection（F2 group）: Immediately after surgery, 0.5 mg flumazenil was administered, followed by 0.3 mg flumazenil 25 minutes later.
  Other Names: Flumazenil at Different Dosages
  Arms: "Flumazenil group 1（F1 group）"+"Flumazenil group 2（F2 group）"
Drug: Saline（C group） — Flumazenil Injection（F2 group）: Immediately after surgery, an equal volume of saline (equal to the volume of 0.5 mg flumazenil) was administered, followed by an equal volume of saline (equal to the volume of 0.3 mg flumazenil) 25 minutes later.
  Other Names: control group
  Arms: Control Group (C group)

SUMMARY:
To investigate the effect of different doses of flumazenil antagonism on remimazolam plasma concentration in patients undergoing renal transplantation under general anesthesia.

DETAILED DESCRIPTION:
During the surgery, other anesthetics, intraoperative monitoring, fluid management, and postoperative pain management were implemented according to a unified standard.

1. Intraoperative Monitoring All study participants underwent the following routine intraoperative monitoring: blood pressure, electrocardiogram, pulse oximetry, end-tidal CO2 pressure, body temperature, and depth of anesthesia monitoring. Additional monitoring such as central venous pressure, invasive continuous arterial blood pressure, and cardiac output was selected based on clinical needs and the attending anesthesiologist's judgment.
2. Anesthetic Regimen

   All study participants underwent general anesthesia with endotracheal intubation and received total intravenous anesthesia with remimazolam. For anesthesia induction, it was recommended to administer remimazolam at a rate of 6-12 mg/kg/h until loss of consciousness; for maintenance, it was recommended to administer at a rate of 0.5-2.0 mg/kg/h. At the end of anesthesia:

   C Group: Immediately after surgery, an equal volume of saline (equal to the volume of 0.5 mg flumazenil) was administered, followed by an equal volume of saline (equal to the volume of 0.3 mg flumazenil) 25 minutes later.

   R1 Group: Immediately after surgery, 0.5 mg flumazenil was administered, followed by an equal volume of saline (equal to the volume of 0.3 mg flumazenil) 25 minutes later.

   R2 Group: Immediately after surgery, 0.5 mg flumazenil was administered, followed by 0.3 mg flumazenil 25 minutes later.

   None of the three groups used inhalation anesthetics such as sevoflurane, or other intravenous sedatives such as midazolam, dexmedetomidine, or etomidate. Intraoperative analgesics were administered with remifentanil via continuous intravenous infusion. Muscle relaxants included cisatracurium, with a single intravenous injection of cisatracurium 0.2 mg/kg for induction to meet muscle relaxation conditions for tracheal intubation, and intermittent single intravenous bolus of cisatracurium 0.05 mg/kg to maintain muscle relaxation as needed for the surgery.
3. Depth of Anesthesia Management Narcotrend was measured as a baseline value within 60 minutes before administration, and intraoperative depth of anesthesia monitoring was conducted using Narcotrend. The dose of remimazolam was adjusted according to hemodynamics to ensure that the patient's anesthesia depth (Narcotrend Index, NCI) was maintained between 27 and 60. (If the NCI value could not be maintained at ≤ 60 or there were signs of potential inadequate anesthesia (e.g., coughing, sweating, and patient movement), and the maximum bolus and infusion doses of remimazolam had been administered, rescue medications such as midazolam or propofol were allowed.)
4. Blood Pressure Management Intraoperative blood pressure control aimed to maintain a mean arterial pressure (MAP) of no less than 65 mmHg, which was the minimum blood pressure tolerated by the anesthesiologist during surgery, not the target value. Higher or lower intraoperative blood pressure management targets could be adopted based on the participant's condition and/or the surgeon's requirements. The use of vasoactive drugs was minimized. If vasoactive drugs were needed, ephedrine 5 mg (maximum dose not exceeding 30 mg) and norepinephrine 10 µg intravenous bolus or continuous infusion were used. Norepinephrine was prepared and used as follows: 2 mg of norepinephrine bitartrate was diluted in 100 mL of saline to a concentration of 20 µg/mL, with an initial dose of 0.01 µg/kg/min. The dose was adjusted in real-time based on intraoperative blood pressure, using the minimum amount of drug necessary to maintain the target MAP. In case of severe bradycardia (<40 beats/min), the norepinephrine infusion rate could be reduced, and an appropriate dose of atropine could be administered intravenously based on the anesthesiologist's judgment.
5. Respiratory Management A lung-protective ventilation strategy was recommended during surgery: setting a tidal volume of 6-8 mL/kg, an inspiratory-expiratory ratio of 1:2, and adjusting positive end-expiratory pressure (PEEP) to 5-10 cmH2O, maintaining end-tidal CO2 pressure between 35-45 mmHg, and using periodic lung recruitment maneuvers. Spontaneous breathing was restored as soon as possible at the end of surgery, and the endotracheal tube was removed.
6. Fluid Management Crystalloids were the primary fluids recommended during surgery, following a moderately liberal fluid management strategy.
7. Other Management Points Comprehensive warming measures were recommended during surgery to maintain core temperature at 37°C. Blood transfusions were recommended based on bleeding and arterial blood gas analysis to maintain hemoglobin levels at ≥70 g/L. Postoperative pain management was selected based on the participant's preoperative preferences and the anesthesiologist's judgment to provide the best pain relief for the participant.
8. Postoperative Management C Group: Immediately after surgery, an equal volume of saline (equal to the volume of 0.5 mg flumazenil) was administered, followed by an equal volume of saline (equal to the volume of 0.3 mg flumazenil) 25 minutes later.

R1 Group: Immediately after surgery, 0.5 mg flumazenil was administered, followed by an equal volume of saline (equal to the volume of 0.3 mg flumazenil) 25 minutes later.

R2 Group: Immediately after surgery, 0.5 mg flumazenil was administered, followed by 0.3 mg flumazenil 25 minutes later.

Arterial blood samples of 3 mL were collected in plastic tubes containing EDTA K3 (Becton Dickinson, Germany) at T1 (end of surgery), T2 (25 minutes after the end of surgery), and T3 (50 minutes after the end of surgery). The arterial catheter was flushed with 2 mL of saline after each sample collection. Samples were kept on ice water and centrifuged at approximately 2000 rpm at 4°C for 10 minutes within 40 minutes of collection. Plasma was separated into polypropylene tubes (Nunc cryogenic vial cryo tubes, Thermo Fisher Scientific, USA) within 15 minutes and stored at -70°C. The sample collection time was recorded. The samples were sent to a third-party testing company for analysis within two months of collection.

Data recorded included the time to eye-opening, extubation time, the amount of remimazolam used, intraoperative analgesic use, hemodynamic parameters at T0 (admission), T1, T2, and T3, MMSE scores 24h and 72h before and after surgery, Narcotrend values at T0, T1, T2, and T3, PACU stay time, and the incidence of nausea and vomiting during PACU stay; postoperative complications such as atelectasis, cardiovascular and cerebrovascular events (stroke, myocardial infarction), all-cause mortality within 30 days postoperatively, total length of hospital stay (days) for survivors within 30 days postoperatively, and unplanned readmissions within 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 65 years
* Patients undergoing elective kidney transplant surgery
* Signed the informed consent for the clinical study

Exclusion Criteria:

* Liver decompensation (Child B/C)
* History of liver transplant
* Previous allergies or other serious adverse reactions to narcotic drugs
* Intraoperative depth monitoring of anesthesia is not expected
* Preoperative ASA rating of 5
* Received general anesthesia in the 30 days prior to surgery or plan to receive it again within 30 days
* Plan to extend airway protection or mechanical ventilation support time after surgery
* Previous participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Remimazolam | T1 (immediately at the end of surgery)
  3ml arterial blood was drawn to determine the blood concentration of remimazolam
Plasma Concentration of Remimazolam | T2 (25 minutes after the end of surgery)
  3ml arterial blood was drawn to determine the blood concentration of remimazolam
Plasma Concentration of Remimazolam | T3 (50 minutes after the end of surgery)
  3ml arterial blood was drawn to determine the blood concentration of remimazolam

SECONDARY OUTCOMES:
Record eye opening time and extubation time | after surgery,an average of 30 minutes
  Record eye opening time and extubation time
remimazolam usage | immediately at the end of surgery
  remimazolam usage
The amount of analgesic drugs used during operation | 3 days after surgery
  The amount of analgesic drugs used during operation
Heart Rate (HR) | T0（Entering the Operating Room, Before Anesthesia）
  Unit: beats per minute (bpm) Measurement of heart rate upon entering the operating room, before anesthesia administration, to monitor baseline cardiac activity.
Blood Pressure (BP) | T0（Entering the Operating Room, Before Anesthesia）
  Unit: millimeters of mercury (mmHg) Measurement of systolic and diastolic blood pressure upon entering the operating room, before anesthesia administration, to monitor baseline blood pressure.
Mean Arterial Pressure (MAP) | T0（Entering the Operating Room, Before Anesthesia）
  Unit: millimeters of mercury (mmHg) Calculation of mean arterial pressure using the formula: (Systolic BP + 2*Diastolic BP) / 3, upon entering the operating room, before anesthesia administration, to monitor baseline arterial pressure.
Oxygen Saturation (SpO2) | T0（Entering the Operating Room, Before Anesthesia）
  Unit: percentage (%) Measurement of blood oxygen saturation upon entering the operating room, before anesthesia administration, to ensure baseline oxygenation levels.
Heart Rate (HR) | T1(immediately at the end of surgery)
  Unit: beats per minute (bpm) Measurement of heart rate upon entering the operating room, before anesthesia administration, to monitor baseline cardiac activity.
Blood Pressure (BP) | T1(immediately at the end of surgery)
  Unit: millimeters of mercury (mmHg) Measurement of systolic and diastolic blood pressure upon entering the operating room, before anesthesia administration, to monitor baseline blood pressure.
Mean Arterial Pressure (MAP) | T1(immediately at the end of surgery)
  Unit: millimeters of mercury (mmHg) Calculation of mean arterial pressure using the formula: (Systolic BP + 2*Diastolic BP) / 3, upon entering the operating room, before anesthesia administration, to monitor baseline arterial pressure.
Oxygen Saturation (SpO2) | T1(immediately at the end of surgery)
  Unit: percentage (%) Measurement of blood oxygen saturation upon entering the operating room, before anesthesia administration, to ensure baseline oxygenation levels.
Heart Rate (HR) | T2（25 minutes after the end of surgery)
  Unit: beats per minute (bpm) Measurement of heart rate upon entering the operating room, before anesthesia administration, to monitor baseline cardiac activity.
Blood Pressure (BP) | T2（25 minutes after the end of surgery)
  Unit: millimeters of mercury (mmHg) Measurement of systolic and diastolic blood pressure upon entering the operating room, before anesthesia administration, to monitor baseline blood pressure.
Mean Arterial Pressure (MAP) | T2（25 minutes after the end of surgery)
  Unit: millimeters of mercury (mmHg) Calculation of mean arterial pressure using the formula: (Systolic BP + 2*Diastolic BP) / 3, upon entering the operating room, before anesthesia administration, to monitor baseline arterial pressure.
Oxygen Saturation (SpO2) | T2（25 minutes after the end of surgery)
  Unit: percentage (%) Measurement of blood oxygen saturation upon entering the operating room, before anesthesia administration, to ensure baseline oxygenation levels.
Heart Rate (HR) | T3（50 minutes after the end of surgery)
  Unit: beats per minute (bpm) Measurement of heart rate upon entering the operating room, before anesthesia administration, to monitor baseline cardiac activity.
Blood Pressure (BP) | T3（50 minutes after the end of surgery)
  Unit: millimeters of mercury (mmHg) Measurement of systolic and diastolic blood pressure upon entering the operating room, before anesthesia administration, to monitor baseline blood pressure.
Mean Arterial Pressure (MAP) | T3（50 minutes after the end of surgery)
  Unit: millimeters of mercury (mmHg) Calculation of mean arterial pressure using the formula: (Systolic BP + 2*Diastolic BP) / 3, upon entering the operating room, before anesthesia administration, to monitor baseline arterial pressure.
Oxygen Saturation (SpO2) | T3（50 minutes after the end of surgery)
  Unit: percentage (%) Measurement of blood oxygen saturation upon entering the operating room, before anesthesia administration, to ensure baseline oxygenation levels.
Mini-Mental State Examination （MMSE )scores were obtained before, 24h and 72h after surgery | Entering the Operating Room, Before Anesthesia
  Scale Description: The MMSE is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language, and visual-spatial skills.
  Unit: Score (0-30) Score Range: The MMSE score ranges from 0 to 30.
  Interpretation of Scores:
  Higher Scores: Indicate better cognitive function. Lower Scores: Indicate worse cognitive function.
  Score Interpretation:
  Cognitive Impairment:
  The maximum score is 30 points. A score of 27-30 points is considered normal, while a score of <27 points indicates cognitive impairment.
  Dementia Classification Criteria:
  Illiterate: ≤17 points Primary School Level: ≤20 points Secondary School Level (including technical secondary school): ≤22 points University Level (including junior college): ≤23 points
  Dementia Severity Grading:
  Mild: MMSE ≥21 points Moderate: MMSE 10-20 points Severe: MMSE ≤9 points
  Data Collection Points:
  Before Surgery (Entering the Operating Room, Before Anesthesia)
Mini-Mental State Examination （MMSE ）scores | 24h after the end of surgery
  Scale Description: The MMSE is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language, and visual-spatial skills.
  Unit: Score (0-30) Score Range: The MMSE score ranges from 0 to 30.
  Interpretation of Scores:
  Higher Scores: Indicate better cognitive function. Lower Scores: Indicate worse cognitive function.
  Score Interpretation:
  Cognitive Impairment:
  The maximum score is 30 points. A score of 27-30 points is considered normal, while a score of <27 points indicates cognitive impairment.
  Dementia Classification Criteria:
  Illiterate: ≤17 points Primary School Level: ≤20 points Secondary School Level (including technical secondary school): ≤22 points University Level (including junior college): ≤23 points
  Dementia Severity Grading:
  Mild: MMSE ≥21 points Moderate: MMSE 10-20 points Severe: MMSE ≤9 points
  Data Collection Points:
  24 Hours After Surgery
Mini-Mental State Examination （MMSE ）scores | 72 h after the end of surgery
  Scale Description: The MMSE is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language, and visual-spatial skills.
  Unit: Score (0-30) Score Range: The MMSE score ranges from 0 to 30.
  Interpretation of Scores:
  Higher Scores: Indicate better cognitive function. Lower Scores: Indicate worse cognitive function.
  Score Interpretation:
  Cognitive Impairment:
  The maximum score is 30 points. A score of 27-30 points is considered normal, while a score of <27 points indicates cognitive impairment.
  Dementia Classification Criteria:
  Illiterate: ≤17 points Primary School Level: ≤20 points Secondary School Level (including technical secondary school): ≤22 points University Level (including junior college): ≤23 points
  Dementia Severity Grading:
  Mild: MMSE ≥21 points Moderate: MMSE 10-20 points Severe: MMSE ≤9 points
  Data Collection Points:
  72 Hours After Surgery
Bispectral Index (BIS) | T0（Entering the Operating Room, Before Anesthesia）
  This outcome measure will record and report the Bispectral Index (BIS) values. The BIS values are quantitative electroencephalographic (EEG) parameters used to assess the depth of anesthesia and sedation levels.
  Bispectral Index (BIS): A value ranging from 0 to 100, where lower values indicate deeper anesthesia and higher values indicate lighter sedation or wakefulness.
Bispectral Index (BIS) | T1(immediately at the end of surgery)
  This outcome measure will record and report the Bispectral Index (BIS) values. The BIS values are quantitative electroencephalographic (EEG) parameters used to assess the depth of anesthesia and sedation levels.
  Bispectral Index (BIS): A value ranging from 0 to 100, where lower values indicate deeper anesthesia and higher values indicate lighter sedation or wakefulness.
Bispectral Index (BIS) | T2（25 minutes after the end of surgery)
  This outcome measure will record and report the Bispectral Index (BIS) values. The BIS values are quantitative electroencephalographic (EEG) parameters used to assess the depth of anesthesia and sedation levels.
  Bispectral Index (BIS): A value ranging from 0 to 100, where lower values indicate deeper anesthesia and higher values indicate lighter sedation or wakefulness.
Bispectral Index (BIS) | T3 (50 minutes after the end of surgery)
  This outcome measure will record and report the Bispectral Index (BIS) values. The BIS values are quantitative electroencephalographic (EEG) parameters used to assess the depth of anesthesia and sedation levels.
  Bispectral Index (BIS): A value ranging from 0 to 100, where lower values indicate deeper anesthesia and higher values indicate lighter sedation or wakefulness.
Duration of Post-Anesthesia Care Unit (PACU) Stay | Before Leaving PACU Post-Surgery
  Unit: Hours The total time spent in the Post-Anesthesia Care Unit (PACU) from the end of surgery until discharge to the ward.
Occurrence of nausea | 3 days after surgery
  Unit: Incidence (Yes/No) The occurrence of nausea during the stay in the PACU, recorded as a binary outcome (Yes or No).
Occurrence of vomiting | 3 days after surgery
  Unit: Incidence (Yes/No) The occurrence of vomiting during the stay in the PACU, recorded as a binary outcome (Yes or No).
Number of Participants with Postoperative Pulmonary Atelectasis, Cardiovascular and Cerebrovascular Adverse Events | 30 days after surgery
  This measure will report the number of participants who experience postoperative pulmonary atelectasis and adverse cardiovascular and cerebrovascular events, including cerebral infarction, cerebral hemorrhage, and heart infarction, within 30 days after surgery.
All-cause death within 30 days after surgery | 30 days after surgery
  All-cause death within 30 days after surgery
Total hospital stay for survivors 30 days after surgery | 30 days after surgery
  Total hospital stay for survivors 30 days after surgery
Unplanned second hospital admission within 30 days after surgery | 30 days after surgery
  Unplanned second hospital admission within 30 days after surgery